CLINICAL TRIAL: NCT02182479
Title: Comparison of the Safety and Efficacy of Berodual® Administered Via Respimat® Device (50 µg Fenoterol Hydrobromide/20 µg Ipratropium Bromide and 25 µg Fenoterol Hydrobromide/10 µg Ipratropium Bromide, 1 Puff q.i.d.) With That Administered Via the MDI (50 µg Fenoterol Hydrobromide/21 µg Ipratropium Bromide, 2 Puffs q.i.d.) in Asthma Patients Over a 12-week Period
Brief Title: Safety and Efficacy of Berodual® Respimat® Compared to Berodual® MDI (Metered Dose Inhaler) in Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215.1104
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (5):
- Berodual® via Respimat®, high dose (Experimental)
  Interventions: Drug: Berodual® via Respimat®, high dose
- Berodual® via Respimat®, low dose (Experimental)
  Interventions: Drug: Berodual® via Respimat®, low dose
- Berodual® via MDI, high dose (Active Comparator)
  Interventions: Drug: Berodual® via MDI, high dose
- Placebo via Respimat® (Placebo Comparator)
  Interventions: Drug: Placebo Respimat®
- Placebo via MDI (Placebo Comparator)
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: Berodual® via Respimat®, high dose
  Arms: Berodual® via Respimat®, high dose
Drug: Berodual® via Respimat®, low dose
  Arms: Berodual® via Respimat®, low dose
Drug: Berodual® via MDI, high dose
  Arms: Berodual® via MDI, high dose
Drug: Placebo Respimat®
  Arms: Placebo via Respimat®
Drug: Placebo MDI
  Arms: Placebo via MDI

SUMMARY:
Study to demonstrate that at least one of the two doses of Berodual® (50 µg fenoterol hydrobromide/20 µg ipratropium bromide and 25 µg fenoterol hydrobromide/10 µg ipratropium bromide, 1 puff q.i.d.) administered via Respimat® gives a bronchodilator response which is not inferior to that obtained from one dose of Berodual® (50 µg fenoterol hydrobromide/21 µg ipratropium bromide, 2 puffs q.i.d.) administered via MDI and that the safety profile is at least as good in asthma patients treated for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchial asthma according to the ATS (American Thoracic Society)
* Age: 18 - 65 years
* Screening FEV1: 40 - 80 % of predicted normal. Predicted normal values will be based on the guidelines for standardised function testing of the European Community for Coal and Steel
* Airway obstruction reversibility: increase in FEV1 12% from baseline and ≥ 200 ml from baseline at 30 minutes after 2 puffs of Berodual® MDI
* Current non-smoker or ex-smoker (with a smoking history of ≤ 10 pack-years) with cessation of smoking ≥ 1 year prior to the screening visit
* Male or female patients
* Ability to be trained in proper use of MDI and RESPIMAT® devices
* Ability to perform technically satisfactory pulmonary function tests
* No hospital admission for an exacerbation and stable dosage of all pulmonary medication in the last four weeks (except for long acting β2 agonists)
* Willingness and ability to sign informed consent form prior to participation in the trial

Exclusion Criteria:

* Patients with significant disease other than asthma, e.g. history of clinically significant cardiovascular, renal, neurological, hepatic or endocrine dysfunction. A clinically significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or which may influence the results of the study or the ability of the patient to participate in and complete the study
* History of myocardial infarction within the last year
* Tuberculosis with indication for treatment
* History of cancer within the last five years, excluding treated basal cell carcinoma
* Patients who have undergone thoracotomy for pulmonary resection of more than one bullae, or with subsequent impaired thoracic muscle performance leading to unsatisfactory lung function testing
* Current psychiatric disorders
* History of life threatening pulmonary obstruction, cystic fibrosis or bronchiectasis
* An upper or lower respiratory tract infection in the four weeks prior to the screening visit (= Visit 1) or during the 2-week run-in period
* Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion
* Patients with AST/ALT (aspartate amino transferase/alanine amino transferase) (SGOT/SGPT (serum glutamic oxaloacetic transaminase/serum glutamic pyruvic transaminase)) > 200%, bilirubin > 150% (except isolated bilirubin increase due to Gilbert's Syndrome), or creatinine > 125% of the upper limit of the normal range
* Intolerance to aerosolised fenoterol- or ipratropium-containing products, and/or hypersensitivity to any of the MDI ingredients
* Patients using oral corticosteroid medication at unstable (i.e. less than 4 weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg prednisone per day or 20 mg every other day
* Beta-blocker medication
* Patients who have taken an investigational drug one month or six half-lives (whichever is greater) prior to the screening visit
* History of drug abuse and/or alcoholism
* Pregnant or nursing women and women of childbearing potential or less than 2 years postmenopausal, who are not using medically approved means of contraception (oral contraceptives, intra-uterine devices or surgical Sterilisation)
* Previous participation in this study
* Patients who need more than 8 puffs of salbutamol (100 µg per puff) rescue medication on 3 or more consecutive days during the run-in period
* Severe bronchial asthma with frequent nocturnal asthma attacks or acute exacerbations induced by recurrent bronchial infections several times per year
* Patients with known hypersensitivity to anticholinergic drugs
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients who did not fill in at least 80% of the diary in the run-in period for both, medication taken and peak expiratory flow rate (PEFR) measurements are considered not compliant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 1998-04; Primary Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Change in average FEV1 (Forced expiratory volume in one second) (AUC0-6 (Area under the curve)) | Pre-dose and 5, 15, 30, 60, 90, 120, 180, 240, 300, 360 minutes post-dose on day 1, 29, 57 and 85

SECONDARY OUTCOMES:
FEV1max | Pre-dose and 5, 15, 30, 60, 90, 120, 180, 240, 300, 360 minutes post-dose on day 1, 29, 57 and 85
Time to onset of therapeutic response | Days 1, 29, 57 and 85
Duration of therapeutic response | Days 1, 29, 57 and 85
Time to peak FEV1 | Pre-dose and 5, 15, 30, 60, 90, 120, 180, 240, 300, 360 minutes post-dose on days 1, 29, 57 and 85
Change in averaged weekly morning and evening pre-dose PEFR (peak expiratory flow rate) | up to day 85
Extent of use of rescue medication | up to day 85
Change in night-time and daytime symptom scores | up to day 85
Overall incidence of adverse events | up to day 85
Number of patients with clinically significant changes in Heart rate | Pre-dose and 15, 30, 60, 90, 120, 180, 240, 300, 360 minutes post-dose on days 1, 29, 57 and 85
Number of patients with clinically significant changes in Blood pressure | Pre-dose and 15, 30, 60, 90, 120, 180, 240, 300, 360 minutes post-dose on days 1, 29, 57 and 85
Number of patients with clinically significant changes from baseline in laboratory investigations | Baseline and day 85
Incidence of paradoxical bronchoconstriction | up to day 85